CLINICAL TRIAL: NCT03677921
Title: A Clinical Trial of Bio-Germanium for the Evaluation of Efficacy on Immune Function Enhancement and Immune Cell Activation
Brief Title: A Clinical Trial of Bio-Germanium for the Evaluation of Efficacy on Immune Function
Acronym: NYG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: YG_immune
Record Dates: First submitted 2018-09-12; First posted 2018-09-19 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Normal Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Group- Bio-Germanium (Experimental): * Ingredient: Bio-Germanium
  * Type: HPMC capsule
  * Weight: 300mg/capsule
  * Directions: 2 capsules, twice a day (1.2g/day of Bio-Germanium)
  * Duration of use: 8 weeks
  Interventions: Dietary Supplement: Investigational Product (Bio-Germanium)
- Control Group - Placebo Product (Placebo Comparator): * Ingredient: Corn starch
  * Type: HPMC capsule
  * Weight: 300mg/capsule
  * Directions: 2 capsules, twice a day
  * Duration of use: 8 weeks
  Interventions: Dietary Supplement: Control Group - Placebo Product

INTERVENTIONS:
Dietary Supplement: Investigational Product (Bio-Germanium) — * Ingredient: Bio-Germanium
  * Type: HPMC capsule
  * Weight: 300mg/capsule
  * Directions: 2 capsules, twice a day (1.2g/day of Bio-Germanium)
  * Storage: Room temperature (below 25℃)
  * Duration of use: 8 weeks
  Arms: Investigational Group- Bio-Germanium
Dietary Supplement: Control Group - Placebo Product — * Ingredient: Corn starch
  * Type: HPMC capsule
  * Weight: 300mg/capsule
  * Directions: 2 capsules, twice a day
  * Storage: Room temperature (below 25℃)
  * Duration of use: 8 weeks
  Arms: Control Group - Placebo Product

SUMMARY:
This study is a 8-week, randomized, double-blind, placebo-controlled clinical trial of Bio-Germanium for the evaluation of efficacy on immune function and immune cell activation.

DETAILED DESCRIPTION:
This study will evaluate Bio-Germanium's efficacy on immune function and immune cell activation in healthy volunteers by assessing improvements in certain immune indices (i.e. NK cell activity, WBC, IFN-γ, TNF-α, IgG1, IgG2, IgM, IL-2, 6, 12).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female volunteers between the ages of 25 to 75 years
2. Screening result for WBC counts in between 4,000 cells/ul and 8,000 cells/ul
3. Volunteers who have agreed to participate in the study and provided a written content by him/herself or through its legal representative

Exclusion Criteria:

1. Those under the treatment for clinically significant acute or chronic diseases in cardiovascular, immune, respiratory, liver, biliary, renal, urinary, nervous, musculoskeletal system as well as psychiatric, infectious, hematologic and neoplastic diseases (exceptions can be made under the discretion of the researcher)
2. Those with uncontrolled hypertension (140/90mmHg or higher, measured after 10 minutes of resting)
3. Those with uncontrolled diabetes (fasting blood glucose levels greater than 126mg/dl or those starting diabetes medication within 3 months)
4. Those received vaccination within 3 months before screening
5. Those with blood AST(GOT) or ALT(GPT) levels greater than 120IU/L
6. Those with blood creatinine level greater than 2.4mg/dL for male and 1.8mg/dL for female
7. Those who have consumed within 2 weeks before screening or are currently consuming health supplements that can affect immune function
8. Those under the severe gastrointestinal symptoms such as heartburn, indigestion, and such
9. Those who are pregnant, breastfeeding or planning to become pregnant during this study
10. Those who are oversensitive or allergic to the investigational product
11. Those who plan to participate in other researches during this study
12. Those who participated in other researches within 4 weeks of the start of this study
13. Those who are deemed inappropriate by the researcher

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-12-10 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
WBC(White blood cell) Count | at 8 week
  WBC(White blood cell) Count
NK(Natural killer) cell activity | at 8 week
  NK(Natural killer) cell activity
Immune related indicator (IFN-γ, IL-2, 6, 12, TNF-α, IgG1, IgG2, IgM) | at 8 week
  Immune related indicator (IFN-γ, IL-2, 6, 12, TNF-α, IgG1, IgG2, IgM)
Evaluation of improvement by the subjects themselves | at 8 week
  Evaluation of improvement by the subjects themselves (Excellent, Good, Unchanged, Worsening, Very aggravated / 5 Step)

SECONDARY OUTCOMES:
Adverse reactions | at 8 week
  Number of Participants with Adverse reactions
Body temperature | at 8 week
  Body temperature

CONTACTS AND LOCATIONS:
Overall Officials: JONGHO LEE, Ph.D., Principal Investigator — Yonsei University
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Yonsei University., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho JM, Chae J, Jeong SR, Moon MJ, Shin DY, Lee JH. Immune activation of Bio-Germanium in a randomized, double-blind, placebo-controlled clinical trial with 130 human subjects: Therapeutic opportunities from new insights. PLoS One. 2020 Oct 19;15(10):e0240358. doi: 10.1371/journal.pone.0240358. eCollection 2020. PMID 33075061